CLINICAL TRIAL: NCT02073942
Title: Cologne Register of Wearable Defibrillator (CRWD)
Status: Completed | Type: Observational
Sponsor: University of Cologne (Other)
Collaborators: Zoll Medical Corporation (Industry)
Responsible Party: Principal Investigator, Guido Michels, PD Dr., University of Cologne
Other Study IDs: 14-050
Record Dates: First submitted 2014-02-24; First posted 2014-02-28 (Estimated); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Myocardial Infarction; Ventricular Dysfunction; Myocarditis
MeSH Terms: conditions — Myocardial Infarction; Ventricular Dysfunction; Myocarditis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month

SUMMARY:
The wearable cardiac defibrillator (WCD) is an alternative to the implantation of cardioverter defibrillator (ICD) for patients at high risk for sudden cardiac death (mostly bridging therapy). The Cologne register of wearable defibrillator (CRWD) is a prospective register for all patient with an indication of wearable defibrillator.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with an indication for wearable defibrillator

Exclusion Criteria:

* childs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with an indication for wearable defibrillator
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-02; Primary Completion 2017-12-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Number of arrhythmic events and arrhythmic risk factors during bridging therapy with wearable defibrillator | 3 years

SECONDARY OUTCOMES:
Total mortality | 1 months and 3 months
  Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cologne, Cologne, Germany